CLINICAL TRIAL: NCT01094093
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending Single-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 139 in Healthy Subjects and Subjects With Moderate to Severe Psoriasis
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 139 in Healthy Subjects and Subjects With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20080767
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Psoriasis
Keywords: Amgen; AMG 139
MeSH Terms: conditions — Psoriasis | interventions — AMG 139

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Part B (Experimental): Four dose levels of AMG 139 administered as a single dose SC or IV in subjects with moderate-severe psoriasis (Part B).
  Interventions: Drug: AMG 139
- Part A (Experimental): Six dose levels of AMG 139 administered as a single dose SC or IV in healthy volunteers.
  Interventions: Drug: AMG 139

INTERVENTIONS:
Drug: AMG 139 — Six dose levels of AMG 139 administered as a single dose SC or IV in healthy volunteers (Part A) and subjects with moderate-severe psoriasis (Part B).

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AMG 139 following single subcutaneous (SC) or intravenous (IV) dose administration in healthy subjects and subjects with moderate to severe psoriasis (PsO).

ELIGIBILITY:
Inclusion Criteria:

Part A - Healthy Volunteers:

* Healthy male or female of non-reproductive potential subjects between 18 to 45 years-of-age
* Body mass index (BMI) between 18 and 32 kg/m2
* Normal or clinically acceptable physical examination, clinical laboratory values, and ECG
* Additional inclusion criteria apply

Part B - Psoriasis Subjects:

* Male or female of non-reproductive potential subjects with PsO between 18 to 55 years-of-age
* Body mass index (BMI) between 18 and 32 kg/m2
* Normal or clinically acceptable physical examination (PE), clinical laboratory values, and ECG; clinically acceptable PE includes evidence of moderate to severe plaque PsO
* Diagnosis of plaque PsO for at least 6 months
* Moderate to severe plaque PsO defined by:
* A minimum PASI score of ≥ 10
* Psoriasis involving ≥ 10% of the Body Surface Area (BSA)
* Additional inclusion criteria apply

Exclusion Criteria:

Parts A - Healthy Volunteers:

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* Recent or on-going infection(s)
* Underlying condition(s) that predisposes the subject to infections
* History of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers in past 5 years
* Additional exclusion criteria apply

Part B - Psoriasis Subjects:

* History or evidence of a clinically significant disorder (including psychiatric), condition or disease that would pose a risk to subject safety or interfere with the study evaluation, procedures or completion;
* Recent or on-going infection(s)
* Underlying condition(s) that predisposes the subject to infections
* Guttate, pustular, or other non-plaque forms of PsO
* Evidence of skin conditions other than PsO (eg, eczema) that would interfere with evaluations of the effect of investigational product on psoriasis
* History of malignancy of any type, other than in situ cervical cancer or surgically excised non-melanomatous skin cancers in past 5 years
* Additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2010-04-11 (Actual); Primary Completion 2011-07-26 (Actual); Study Completion 2011-07-26 (Actual)

PRIMARY OUTCOMES:
Safety & tolerability: treatment-emergent AEs including clinically significant changes in physical examinations, safety lab tests, ECG, vital signs, or immunogenicity to AMG 139 | 16-24 weeks

SECONDARY OUTCOMES:
Characterization of the pharmacokinetics (PK) of AMG 139 | 16-24 weeks
Psoriasis Activity and Severity Index (PASI) scores (Part B only) | 16-24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Nucleus Network Limited, Melbourne, Victoria
  - Clinical Medical and Analytical eXcellence (CMAX), Adelaide
  - QPharm Pty Limited, Herston
- Auckland Clinical Studies Ltd, Grafton, New Zealand